CLINICAL TRIAL: NCT01087541
Title: SEGUDIAB Study: Safety in Diabetic Patients. Evaluation of an Educational Program for the Professionals to Improve the Safety in Diabetic Patients
Brief Title: SEGUDIAB Study: Evaluation of Safety in the Diabetic Patients
Acronym: SEGUDIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government); Fundación Avedis Donabedian (Unknown)
Responsible Party: Jordi Gol i Gurina Foundation, Jordi Gol i Gurina Foundation
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SEGUDIAB
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Results first posted 2011-03-24 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus
Keywords: Patient's Safety; Diabetes mellitus; Public Health for professionals; Safety; Public health
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual clinical health care
- Intervention (Experimental): Behavioural program of education for health professionals. Standardized program of 6 hours for health professionals ( doctors and nurses )
  Interventions: Behavioral: Educational program 6-hour standardized

INTERVENTIONS:
Behavioral: Educational program 6-hour standardized — 6-hour standardized program for adults ( doctors and nurses )
  Other Names: Standardized educational programs; Patients safety
  Arms: Intervention

SUMMARY:
The safety in the diabetic patient refer so much to the accuracy of the treatment and to the handling of the diabetic in security topics. Therefore, is not only an economic question, but a more global concept that means to receive an accurate sanitary attention in line with the available evidences nowadays.

OBJECTIVE: To analyse if a brief intervention educative on the primary care professionals is followed of an improvement in the safety of the diabetic patients.

METHODS: Cluster Clinical trial, completely in primary care, on 10 basic health areas (BHA) with a random distribution of the educative intervention to realize on the sanitary professionals (5 intervention/5 control). The intervention is an educative system on adults, brief (6 hours) but with periodic reminders. To improve his skills and attitudes for the diabetics. The group control follows his usual clinical practice on the diabetics.

The participation was voluntary. The centres have been matched, being comparable in population and other characteristics, except the specific intervention; ranging between the 6-8% the prevalence observed of type 2 diabetes (T2D) in all the cases. Finally, we selected only between 45 until 75 years old as operative age group of the 45 until the 75 years like operative aim.

Inclusion criteria: T2D or T1D with age comprised between 45 and 75 years; recorded in the informatic software for primary care.

Exclusion criteria: serious or terminal illness or patients controlled exclusively by specialists.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetes
* Aged between 45 and 75 years

Exclusion Criteria:

* No data in informatic system
* Severe illness
* Controlled only by specialists

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6830 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Cabré, MD, PhD, Principal Investigator — Catalan Institute of Health
Locations (1):
- Primary Health Care. Catalan Health Institute. Tarragona-Reus, Reus, Tarragona, Spain

REFERENCES:
- [Derived] Cabre JJ, Ripoll M, Hernandez JM, Basora J, Bejarano F, Arija V. Safety during the monitoring of diabetic patients: trial teaching course on health professionals and diabetics - SEGUDIAB study. BMC Public Health. 2011 Jun 5;11:430. doi: 10.1186/1471-2458-11-430. PMID 21639938

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Behavioural program of education for health professionals of the study
- Control Group: Usual healthcare of diabetics patients
Period: Overall Study
Arm/Group | Intervention | Control Group
Started | 3307 | 3523
Completed | 3307 | 3523
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control Group | Total
Number analyzed (Participants) | 3307 | 3523 | 6830
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2987 | 3001 | 5988
  >=65 years | 320 | 522 | 842
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1907 | 2000 | 3907
  Male | 1400 | 1523 | 2923
Region of Enrollment [Number; unit: participants]
  Spain | 3307 | 3523 | 6830

OUTCOME MEASURES:

1. Primary Outcome: Glycosylated Haemoglobin A1c at Start
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Intervention | Control Group
Number analyzed (Participants) | 3307 | 3523
Percentage | 6.64 (1.60) | 6.76 (1.67)

2. Secondary Outcome: BMI ( Body Mass Index ) at Start
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Intervention | Control Group
Number analyzed (Participants) | 3307 | 3523
kg/m2 | 26.9 (9.7) | 27.1 (9.6)

3. Secondary Outcome: BMI at 6 Months
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Intervention | Control Group
Number analyzed (Participants) | 3307 | 3523
kg/m2 | 30.0 (5.2) | 30.1 (5.8)

4. Primary Outcome: Glycosylated Haemoglobin A1c at 6 Months
Description: Glycohemoglobin A1c at 6 months.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Intervention | Control Group
Number analyzed (Participants) | 3307 | 3523
Percentage | 6.81 (1.49) | 7.00 (1.64)
Statistical Analysis 1: Comparison: Intervention vs Control Group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI [0 to 1], Standard Deviation 0.5

5. Secondary Outcome: Blood Pressure ( Systolic / Diastolic )
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Control Group
Number analyzed (Participants) | 3307 | 3523
mmHg
  Systolic | 130.3 (18.5) | 131.5 (18.6)
  Diastolic | 72.6 (11.9) | 73.7 (11.8)

6. Secondary Outcome: Systolic and Diastolic Blood Pressure
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention | Control Group
Number analyzed (Participants) | 3307 | 3523
mmHg
  Systolic | 130.2 (18.4) | 129.9 (19.5)
  Diastolic | 72.9 (10.5) | 76.2 (12.8)
Statistical Analysis 1: Comparison: Intervention vs Control Group; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 5, 95% CI 2-sided [2 to 15], Standard Deviation 5

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious events are death or another event due to the study's protocol. As this is an educational project in professionals, we had been not any serious event.
Groups:
- Intervention Group: Intervention group: educational program
- Control Group: Usual healthcare
Arm/Group | Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/3307 | 0/3523
Other Adverse Events (participants affected / at risk) | 2/52 | 1/87
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=52) | Control Group (N=87)
Drug interactions not serious (Investigations) | 2 (2) | 1 (1) — The assessment for drug interactions was performed by informatic methods. The adverse event was concomitant treatment with gemfibrozil plus glitazones, that is not recommended.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No